CLINICAL TRIAL: NCT04890106
Title: A Randomized ( 1:1), Double-Masked, Multi-Center, Two-Treatment, Single-Period, Parallel Design, Mutiple Dose Bioequivalence Study With Clinical End-Point of Bimatoprost Ophthalmic Solution 0.01% of Mankind Pharma Limited With LUMIGAN (Bimatoprost Ophthalmic Solution) 0.01% of Allergan, Inc., in Subjects With Chronic Open-Angle Glaucoma Or Ocular Hypertension in Both Eyes
Brief Title: Bioequivalence Study With Clinical Endpoint Comparing Bimatoprost Ophthalmic Solution 0.01% to LUMIGAN® In The Treatment of Chronic Open-Angle Glaucoma
Acronym: Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mankind Pharma Limited (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCC/2021/004
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Ophthalmic Solutions; Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost 0.01% Ophthalmic Solution (Experimental): Bimatoprost Pharmaceutical dosage form: Ophthalmic Solution Strength: 0.01% Manufactured by: Mankind Pharma Limited, India.
  Intervention Drug: Test - Bimatoprost 0.01% Ophthalmic Solution
  Interventions: Drug: Test - Bimatoprost 0.01% Ophthalmic Solution
- LUMIGAN® 0.01% Ophthalmic Solution (Active Comparator): LUMIGAN® ( Contains Bimatoprost) Pharmaceutical dosage form: Ophthalmic Solution Strength: 0.01% Manufactured by: Allergan, Inc.,
  Intervention Drug: Reference - Bimatoprost 0.01% Ophthalmic Solution
  Interventions: Drug: Reference - LUMIGAN® (Bimatoprost 0.01% Ophthalmic Solution)

INTERVENTIONS:
Drug: Test - Bimatoprost 0.01% Ophthalmic Solution — Subjects in one arm will receive one drop of the test drug in both the eyes every evening at approximately 10:00 pm ± 2 hours for 42 days.
  Arms: Bimatoprost 0.01% Ophthalmic Solution
Drug: Reference - LUMIGAN® (Bimatoprost 0.01% Ophthalmic Solution) — Subjects in the second arm will receive one drop of the reference drug in both the eyes every evening at approximately 10:00 pm ± 2 hours for 42 days.
  Arms: LUMIGAN® 0.01% Ophthalmic Solution

SUMMARY:
This is a randomized, double-masked, two-treatment, single-period, parallel design, multiple dose at multiple clinical trial sites designed to demonstrate bioequivalence with clinical endpoint in subjects with chronic open-angle glaucoma or ocular hypertension in both eyes.

Test Product - Bimatoprost Ophthalmic Solution, 0.01% of Mankind Pharma Limited, India

Reference Product - LUMIGAN® (Bimatoprost Ophthalmic Solution) 0.01% of Allergan, Inc.,

DETAILED DESCRIPTION:
Subjects with chronic open-angle glaucoma or ocular hypertension in both the eyes and meeting all the mentioned inclusion criteria and none of the exclusion criteria will be identified. Qualifying Intra Ocular Pressure (IOPs) following wash-out, at baseline (Day 0 at anytime of the day) should be ≥ 22 milli meter mercury (mm Hg) and ≤ 34 mm Hg in each eye and any asymmetry of IOP between the eyes no greater than 5 mm Hg.

Subjects will receive one drop of investigational product (either A or B) in both the eyes every evening at approximately 10:00 pm ± 2 hours for 42 days.

The study subjects will undergo clinical evaluations throughout the study in order to assess efficacy and safety. Study subject primary endpoint evaluation will be assessed after 2 weeks (day 14) and 6 weeks ( Day 42) of treatment for each study subject deemed eligible for evaluation.

The primary bioequivalence comparison is between the test and reference products for the mean difference in intraocular pressure (IOP) of both eyes between the two treatment groups at six time points, i.e., at 00.00 hours (between 8:00am and 10:00 am), 04.00 hours (at 4 hours after 00.00 hours) and 08.00 hours ( at 8 hours after 00.00 hours) on Day 14 (week 2) and Day 42 (week 6) visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to provide voluntary informed consent and to follow the protocol requirements
2. Male or non-pregnant females aged ≥18 years having body mass index (BMI) ≥ 17 calculated as weight in kg/height in m2.
3. Subjects with chronic open-angle glaucoma or ocular hypertension in both eyes.
4. Subjects requiring treatment of both the eyes and can discontinue use of all ocular hypotensive medication(s) or switch ocular hypotensive medications and undergo an appropriate washout period
5. Adequate wash-out period prior to baseline of any ocular hypotensive medication as per the table below (In order to minimize potential risk to subjects due to intraocular pressure (IOP) elevations during the washout period, the investigator may choose to substitute a parasympathomimetic or carbonic anhydrase inhibitor in place of a sympathomimetic, alpha-agonist, beta-adrenergic blocking agent, or prostaglandin; however, all subjects must have discontinued all ocular hypotensive medications for the minimum washout period
6. Baseline (Day 0/hour 0) IOP ≥ 22 mm Hg and ≤ 34 mm Hg in each eye and difference in IOP between the eyes is not greater than 5 mm Hg
7. Subject's IOP is likely to be controlled with monotherapy as per the discretion of the investigator
8. Baseline best-corrected visual acuity equivalent to 20/200 (6/60) or better in each eye
9. Women of child-bearing potential (defined as women physiologically capable of becoming pregnant, unless they are using an effective contraception method during dosing of the investigational product) practicing any two acceptable contraception methods

   Acceptable methods of contraception are:
   1. Oral or parenteral (injection) , patch, or implant) hormonal contraception which has been used continuously for at least one month prior to the first dose of study medication
   2. Intrauterine device (IUD) or intrauterine system IUS)
   3. A double barrier method of contraception (Condom and occlusive cap or condom and spermicidal agent)
   4. Male sterilization (at least six months prior to the screening, should be the sole male partner for that subject)
   5. Female sterilization (surgical bilateral oophorectomy) or tubal ligation at least six weeks prior to study participation
   6. Total abstinence, partial abstinence is not acceptable
10. No history of addiction to any recreational drug or drug dependence or alcohol addiction

Exclusion Criteria:

1. Hypersensitivity to Bimatoprost or related class of drugs or any of the excipients of the formulation
2. Severe hepatic or renal impairment
3. Current or history within two months prior to the baseline of any other significant ocular disease, e.g., corneal edema, uveitis, ocular infection, or ocular trauma in either eye. Note: - Stable myopia, strabismus and cataracts (as per investigator's discretion) will be allowed provided other inclusion/exclusion criteria are met
4. Current corneal abnormalities that would prevent accurate IOP readings with the Goldmann applanation tonometer
5. Functionally significant visual field loss
6. Use of an intraocular corticosteroid implant at any time prior to the baseline
7. Use of contact lens within one week prior to the baseline
8. Use of 1) topical ophthalmic corticosteroid, or 2) topical corticosteroid within two weeks prior to the baseline
9. Use of 1) systemic corticosteroid or 2) high-dose salicylate therapy defined as 325mg/day taken on three consecutive days, within one month prior to the baseline
10. Use of intravitreal or subtenon injection of ophthalmic corticosteroid within six months prior to the baseline
11. Underwent any other intraocular surgery (e.g., cataract surgery) within six months prior to the baseline
12. Underwent refractive surgery, filtering surgery, or laser surgery for IOP reduction (e.g., laser trabeculoplasty) within twelve months prior to the baseline
13. Amblyopia/only one sighted eye
14. Subjects with a past history of IOP previously uncontrolled on bimatoprost monotherapy
15. Severe retinal disease or other severe ocular pathology, such as glaucomatous damage with a cup/disk ratio greater than 0.8, split fixation, or functionally significant (in the investigators' opinion) visual field loss
16. Chronic use of any systemic medication that may affect IOP with less than a three-month stable dosing regimen (i.e., sympathomimetic agents, beta-adrenergic blocking agents, alpha agonists, alpha-adrenergic blocking agents, calcium channel blockers, angiotensin-converting enzyme inhibitors, etc.)
17. Known history or presence of any uncontrolled systemic disease (e.g., cardiovascular disease, hypertension, diabetes mellitus, hepatic impairment, etc.)
18. History of recurrent ocular seasonal allergies within the past two years
19. Any other medical condition or severe intercurrent illness that, in the investigator's opinion, may make it undesirable for the subjects to participate in the study and would limit adherence to the study's requirements
20. Pregnant or lactating woman
21. Subjects with suspected signs and symptoms of COVID-19/confirmed novel coronavirus infection (COVID-19) or with a recent history (within 14 days) of travel/contact with any COVID-19 positive subject/isolation/quarantine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Mean Difference in Intraocular Pressure (IOP) of Both Eyes Between the Two Treatment Groups at Six Time Points | Day 14 and 42 at 00.00 hours (between 8:00 AM and 10:00 AM), 04.00 hours (at 4 hours after 00.00 hours), and 08.00 hours (at 8 hours after 00.00 hours)
  Change in mean difference in intraocular pressure (IOP) of both the eyes between the two treatment groups at six time points, i.e., at 00.00 hours (between 8:00 am and 10:00 am), 04.00 hours (at 4 hours after 00.00 hours), and 08.00 hours (at 8 hours after 00.00 hours) on Day 14 (week 2) and Day 42 (week 6) visits.

SECONDARY OUTCOMES:
Safety and efficacy of Bimatoprost 0.01% Ophthalmic Solution | Safety will be evaluated throughout the study (6 weeks) and telephonic safety follow-up on day 49±3 days
  To monitor the adverse events and safety of the subjects and tolerability of Bimatoprost 0.01% Ophthalmic Solution

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - CBCC Global Research Site:011, Bakersfield, California
  - CBCC Global Research Site 016, Mission Hills, California
  - CBCC Global Research Site 017, Newport Beach, California
  - CBCC Global Research Site: 012, Newport Beach, California
  - CBCC Global Research Site 013, Pasadena, California
  - CBCC Global Research Site 019, Petaluma, California
  - CBCC Global Research Site 015, San Diego, California
  - CBCC Global Research Site 020, Pembroke Pines, Florida
  - CBCC Global Research Site 018, Houston, Texas